CLINICAL TRIAL: NCT03395145
Title: Valuation of Bone Volume Changes After Socket Preservation Using Geistlich Bio-Oss® Collagen and Geistlich Mucograft® Seal Compared to Natural Healing After Tooth Extraction
Brief Title: Bone Volume Changes After Socket Preservation Using Geistlich Bio-Oss Collagen and Mucograft Seal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0507-17-RMB CTIL
Record Dates: First submitted 2018-01-01; First posted 2018-01-10 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Bio-Oss; Mucograft

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-Oss Collagen and Mucograft Seal (Experimental): Bone volume Changes after socket preservation using Geistlich Bio-Oss® Collagen and Geistlich Mucograft® Seal
  Interventions: Device: Geistlich Bio-Oss® Collagen and Geistlich Mucograft® Seal
- Natural healing (No Intervention): Evaluation of Bone volume Changes after tooth extraction (natural healing)

INTERVENTIONS:
Device: Geistlich Bio-Oss® Collagen and Geistlich Mucograft® Seal — Geistlich Bio-Oss® Collagen is intended to be used for filling bone defects and for bone augmentation after tooth extraction
  Arms: Bio-Oss Collagen and Mucograft Seal

SUMMARY:
Evaluation of Bone volume Changes after socket preservation using Geistlich Bio-Oss® Collagen and Geistlich Mucograft® Seal compared to natural healing after tooth extraction

DETAILED DESCRIPTION:
In the last decade dental implants have become widely used for oral rehabilitation. But, the usage of dental Implants might be difficult in cases of alveolar bone deficiencies.

Different ridge preservation techniques were successfully used, using membrane with or without bone substitutes.new grafting material is Mucograft Seal, a collagen matrix graft, which originally used as an alternative to the connective tissue graft for the treatment of gingival recessions. Mucograft has demonstrated a good tissue reaction with high biocompatibility and a low shrinkage tendency, in order to increase the amount of keratinized gingiva in the augmented area.

Study Hypothesis: The observed changes in ridge dimensions when using Geistlich Bio-Oss® Collagen and Geistlich Mucograft® Seal as ridge preservation will be less pronounced in comparison to natural healing after tooth extraction.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Patients of 18 years or older.
* Patients in need of a tooth extraction in the area of premolars, canines or incisors due to periodontal and/or dental reasons, provided that the socket walls are intact (bone dehiscence of max. 4mm limited to one bone wall).
* Patients who need implant placement at the site of extraction.

Exclusion Criteria:

* Inability to complete or understand the informed consent process.
* Bone dehiscence at extraction socket of more than 4 mm or 4 mm at more than one bony wall.
* Pregnant or lactating women.
* Patients who use medications that affect bone metabolism such as IV bisphosphonates.
* Heavy smokers (more than 10 cigarettes per day).
* Patients with removable prosthesis, which might compress the treated site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-27 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2022-07-17 (Actual)

PRIMARY OUTCOMES:
socket width mm | baseline (prior to tooth extraction) and 6 months (implant placement) and at 21 month (one year after loading
  The socket width (buccal-lingual aspect) will be assessed at the following reference points:
  1. 3-(∆ACH pre-post) millimeters apical to the alveolar crest, where the buccal and lingual walls are intact.
  2. 5-(∆ACH pre-post) millimeters apical to the alveolar crest, where the buccal and lingual walls are intact.
  3. The width of each cortical buccal and lingual bone plate, 3 millimeters apical to the alveolar crest.
  4. The width of each cortical buccal and lingual bone plate, 5 millimeters apical to the alveolar crest.
alveolar height mm | baseline (prior to tooth extraction) and 6 months (implant placement) and at 21 month (one year after loading
  Alveolar crest height (ACH) will be measured from the apical part of the stent to the bone crest at the mid M-D distance of the socket.
keratinized tissue mm | baseline (prior to tooth extraction) and 6 months (implant placement) and at 21 month (one year after loading
  In the lower jaw the keratinized tissue width will be measured from the apical part of the stent to the mucogingival line on the buccal and lingual sides. On the upper jaw only the keratinized tissue on the buccal side will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Machtei, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Dept. of Periodontology, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No